CLINICAL TRIAL: NCT02564679
Title: Effects of Sleeve Gastrectomy on Hepatic and Metabolic Abnormalities in Adolescents With Complicated Morbid Obesity and NAFLD
Brief Title: Sleeve Gastrectomy in Adolescents With Complicated Morbid Obesity and NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Valerio Nobili, Professor, Chief of Hepatometabolic Department, Bambino Gesù Hospital and Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LSG_metabolic profile
Record Dates: First submitted 2015-09-23; First posted 2015-10-01 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Morbid Obesity; NAFLD
Keywords: bariatric surgery; sleeve gastrectomy
MeSH Terms: conditions — Obesity, Morbid; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleeve gastrectomy (Experimental): These patients are surgically treated with laparoscopic sleeve gastrectomy in association to lifestyle intervention (hypocaloric diet and physical activity)
  Interventions: Procedure: Laparoscopic Sleeve gastrectomy (LSG)
- Lifestyle Intervention (Experimental): These patients are treated with lifestyle intervention (hypocaloric diet and physical activity)
  Interventions: Behavioral: Lifestyle Intervention

INTERVENTIONS:
Procedure: Laparoscopic Sleeve gastrectomy (LSG) — These patients (no. 20) are assessed by clinical and psychological evaluation (auxological parameters, blood pressure and personal and family history), blood tests (liver function test's (LFT's), uric acid, lipid and gluco-insulinemic profile with oral glucose tolerance test (OGTT)), abdominal ultrasound at time of enrollment.
  They are treated with laparoscopic sleeve gastrectomy associated to lifestyle intervention. Concomitantly to surgical intervention, liver biopsy is performed.
  At 6 and 12 months after LSG the patients are evaluated with laboratory, clinical and echographic assessment. Moreover, one year after LSG liver biopsy is repeated.
  Arms: Sleeve gastrectomy
Behavioral: Lifestyle Intervention — These patients (no. 20) are assessed by clinical and psychological evaluation (auxological parameters, blood pressure and personal and family history), blood tests (liver function test's (LFT's), uric acid, lipid and gluco-insulinemic profile with oral glucose tolerance test (OGTT)), abdominal ultrasound at time of enrollment.
  They are treated with lifestyle intervention. At 6 and 12 months after enrollment the patients are evaluated with laboratory, clinical and echographic assessment.
  Arms: Lifestyle Intervention

SUMMARY:
Pediatric obesity has become a critical health problem worldwide, increasing the premature onset of obesity-related morbidities. This phenomenon has induce an increase in the incidence of serious health complications starting in childhood and adolescence. Lifestyle interventions, including diet and regular physical activity, are the cornerstone of current medical management. Unfortunately, these interventions are often ineffective in providing a meaningful and long-lasting weight loss necessary to change health outcomes. It has been demonstrated that an early intervention in obesity in children and adolescents, inducing weight loss by performing bariatric surgery in carefully selected patients, can dramatically reduce the risk of adulthood obesity and obesity-related diseases, including non-alcoholic fatty liver disease (NAFLD).

Recent evidence suggest that bariatric surgery can improve metabolic complications and liver involvement in patients affected by morbid obesity.

ELIGIBILITY:
Inclusion criteria:

* BMI>40 kg/m2 with severe comorbidities
* Type 2 diabetes mellitus
* Moderate-to-severe sleep apnea
* Pseudotumor cerebri
* NASH with advanced fibrosis (ISHAK score>1)
* BMI>50 kg/m2 with mild comorbidities
* Hypertension
* Dyslipidemia
* Mild obstructive sleep apnea
* Chronic venous insufficiency
* Panniculitis
* Urinary incontinence
* Impairment in activities of daily living
* NASH
* Gastroesophageal reflux disease
* Severe psychological distress
* Arthropathies related to weight

Exclusion Criteria:

* Documented substance abuse problem
* Medically correctable cause of obesity
* Disability that would impair adherence to postoperative treatment, present pregnancy, or breast-feeding

The patients included in the present study were enrolled according to the recent indications for bariatric surgery in severly obese adolescents of Hepatology Committee of European Society of Pediatric Gastroenterology, Hepatology And Nutrition (ESPGHAN) (JPGN 2015;60: 550-561)

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Improvement of metabolic parameters | 12 months
  Improvement of serum levels of cholesterol (mg/dl), triglycerides (mg/dl), HDL (mg/dl), LDL (mg/dl), uric acid (mg/dl), and gluco-insulinemic profile (serum concentration during standard oral glucose tolerance test - OGTT)
Improvement of liver parameters | 12 months
  Improvement of Aspartate aminotransferases (U/L) and Alanine aminotransferases (U/L) serum levels

SECONDARY OUTCOMES:
Improvement of liver histology | 12 months
  improvement of liver histology assessed as Non-alcoholic steatohepatitis score (NAS score) in patients treated with sleeve gastrectomy